CLINICAL TRIAL: NCT01550939
Title: A Single-Center, Open-Label, Randomized Clinical Study Measuring Time Needed for Testing Between the Haag-Streit Lenstar 900 Version i4 and the Carl Zeiss IOL Master 500 Instruments
Brief Title: Time Study for Biometry Measurements With the Lenstar and IntraOcularLens (IOL) Master 500
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haag Streit USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS1 Time Study 2
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Pseudoaphakia
Keywords: Biometry of the Eye; Intraocular Lens Implantation; IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Time Comparison between the Lenstar and IOLMaster (No Intervention)
  Interventions: Device: Ophthalmic Biometer

INTERVENTIONS:
Device: Ophthalmic Biometer — One complete biometry examination
  Other Names: Haag-Streit Lenstar; Zeiss IOL Master 500

SUMMARY:
The objectives of this study are to determine the time needed to complete a full set of measurements (Total Ophthalmic Exam, Subject Data Entry and Acquisition of the Measurement) by each test device, the Lenstar 900 Version i4 and IOL Master 500.

DETAILED DESCRIPTION:
This is an open-label study randomized by sequence. Each eligible subject who signs a consent form and fulfills all Inclusion/Exclusion criteria will undergo ophthalmic measurements by the two test products:

A. Haag-Streit Lenstar Version i4

B. Zeiss IOL Master 500

The order of measurements for the IOL Master 500 and the Haag-Streit Lenstar Version i4 will he randomized. The two possible sequences will be balanced (approximately 22 eyes each: AB,BA). One eye of each subject will be measured. Time needed to complete testing will be measured utilizing a stop-watch. Total time needed to complete all measurements of the study eye using each of the test products to capture a complete ophthalmic exam with the devices standard operating settings set to automatic measurement and analysis will be calculated by the following start and stop points:

First Timed Measurement: Measurement Acquisition Start: When the technician starts to acquire tbe first measurement Stop: When the technician has completed all measurements

Second Timed Measurement: Subject Data Entry Start: When the technician starts to enter the subject data. Stop: When the technician has completed subject data entry.

Third Timed Measurement: Complete Ophthalmic Exam with each test product Start: When tbe subject is seated at the instrument, just prior to the technician entering any subject data into the test product.

Stop: Upon completion of all measurements using one of the test products, just prior to printing results.

Three trained technicians will operate tbe same study devices (Haag-Streit Lenstar Version i4 and IOL Master 500). Approximately equal number of subjects will be assigned to each technician.

ELIGIBILITY:
Inclusion Criteria:

Subjects wbo meet all of the following criteria are eligible to participate in tbe study:

1. Male or female l8 years of age or older on the date of Informed Consent.
2. At least one eye of each subject must be a phakic eye.
3. Subject must be able to fixate on a target.
4. Able to understand and willing to sign tbe informed consent.

Exclusion Criteria:

Subjects will be excluded from the study if the following applies:

1. History of corneal surgery.
2. Use of contact lenses during tbe ophthalmic exam or up to two hours prior to the exam.
3. Any ophthalmic condition preventing use of either of the instruments used in the study.
4. Any ophthalmic condition which might impair tbe validity of results from any of the instruments used in the study.
5. Any medical condition, which, in tbe Investigator's judgment, interferes with the subjects ability to comply with tbe protocol, compromises subject safety, or interferes with tbe interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Time to complete a full examination | At Study Visit (study consists of 1 visit only)
  Time to complete a full ophthalmic exam(as measured from the time of subject placement just prior to the technician completing data entry at the test product, to the beginning of data printing) for each, the IOL Master 500 and the Haag-Streit Lenstar Version i4.

SECONDARY OUTCOMES:
Data Entry Time Measurement | At Study Visit (study consists of 1 visit only)
  Additional Time Measurements - Data Entry from the IOL Master 500 and the Haag-Streit Lenstar Version i4.
Measurement Acquisition Time Measurement | At Study Visit (study consists of 1 visit only)
  Additional Timed Measurements - Measurement Acquisition from the IOL Master 500 and the Haag-Streit Lenstar Version i4.
Adverse Events | Duration of study from signing informed consent to Study Visit (study consists of 1 visit only)
  Any adverse events associated with the test products

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Snyder, MD, Principal Investigator — Cincinnati Eye Institute
Locations (1):
- Cincinnati Eye Institute, Cincinnati, Ohio, United States